CLINICAL TRIAL: NCT03048188
Title: Clinical Application Observation of Manuka Honey in Second- and Grafted Third-degree Burns
Brief Title: Manuka Honey in Second- and Grafted Third-degree Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-265
Record Dates: First submitted 2017-01-28; First posted 2017-02-09 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Second-degree Burn; Third-Degree Burn
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (1):
- Burn with or without split-skin graft (Experimental): Second degree burns and third degree burns with split-skin graft that need wound dressings
  Interventions: Other: wound dressing

INTERVENTIONS:
Other: wound dressing — Manuka honey wound dressing

SUMMARY:
Treatment strategies of II. degree burn wounds and split-skin grafted III. degree burn wounds aim at reducing infection and improving reepithelialization. The aim of this study is to evaluate time to reepithelialization, pain, microbiology and handling of manuka honey dressings with second-degree burn wounds and split-skin grafted burn wounds.

DETAILED DESCRIPTION:
In plastic and reconstructive surgery, treatment strategies of second-degree burn wounds and split-skin grafted third-degree burn wounds aim at reducing infection and improving reepithelialization. Although previous studies indicate that burn patients benefit from wound dressings containing manuka honey, only a few studies can be found. Therefore, the aim of this study is to evaluate time to reepithelialization, pain, microbiology and handling of manuka honey dressings with second-degree burn wounds and split-skin grafted burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Consent-capable male and female patients (or guardian)
* ≥18 years of age
* ability to asses pain

Exclusion Criteria:

* Immunosuppressive Therapy
* Clinical wound infection
* Allergy against honey
* Relationship to someone who is involved in the study design or assessment
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Epithelialization | Up to 1 year
  Rate of Epithelialization in percent

SECONDARY OUTCOMES:
Pain | Up to 1 year
  Visual analog scale (VAS)
Microbiology | Up to 1 year
  Microbiological smear is assessed by gram+, gram- or no bacterium
Handling | Up to 1 year
  Scale (0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University of Lübeck, University Hospital Schleswig-Holstein
Locations (2):
- Germany (2):
  - University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - University of Schleswig-Holstein, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No